CLINICAL TRIAL: NCT06252051
Title: Effectiveness of Trivalent Influenza Vaccine (TIV) in Type 2 Diabetes Mellitus (T2DM) Patients With and Without Complications of Chronic Kidney Disease (CKD): A Clinical Observational Study on Antibody Titers and Dynamic Changes in IL-2 and IL-6 Cytokines
Brief Title: Effectiveness of Trivalent Influenza Vaccine (TIV) in Type 2 Diabetes Mellitus (T2DM) Patients With and Without Complications of Chronic Kidney Disease (CKD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Collaborators: Biofarma (Industry); Universiti Sains Malaysia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S3-202401.01
Record Dates: First submitted 2024-01-28; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Influenza; Vaccine Reaction; Diabetes Mellitus; Chronic Kidney Diseases
Keywords: Immunogenicity; Trivalent Influenza Vaccine; Diabetes Mellitus; Chronic Kidney Diseases
MeSH Terms: conditions — Influenza, Human; Diabetes Mellitus; Renal Insufficiency, Chronic | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trivalent Vaccine (Experimental)
  Interventions: Drug: Trivalent Influenza Vaccine

INTERVENTIONS:
Drug: Trivalent Influenza Vaccine — We divided the participants into three groups: one comprising healthy individuals, another consisting of those with type 2 diabetes mellitus (T2DM), and the last group comprising individuals with T2DM and chronic kidney disease (CKD). All participants will receive a trivalent influenza vaccine, and various parameters will be observed.

SUMMARY:
This study assesses the effectiveness of the seasonal flu vaccine in individuals with Type 2 Diabetes Mellitus (T2DM) with and without Chronic Kidney Disease (CKD), as well as in healthy individuals. Additionally, the study investigates the dynamics of cytokines, specifically IL-2 and IL-6, in the three groups following influenza vaccination. The findings from these studies will contribute to our understanding of the safety and efficacy of the influenza vaccine in T2DM and T2DM-CKD, shedding light on inflammation changes and informing future research on mitigation strategies.

DETAILED DESCRIPTION:
The aim of this study is to assess the effectiveness of the influenza vaccine in the T2DM group, T2DM-CKD group, and healthy individuals without DM or CKD as a comparison. Patients with T2DM are characterized by low-grade inflammation, making them susceptible to infections, particularly influenza, leading to increased ICU admissions and mortality rates. Diabetes mellitus is also a major cause of declining kidney function, with complications known as diabetic kidney disease, ultimately progressing to chronic kidney disease, the most common cause of patients undergoing haemodialysis. The vulnerability to influenza infections prompts the recommendation for influenza vaccination in T2DM patients. Chronic kidney disease is a complication of diabetes that becomes intriguing to study regarding the effectiveness of the influenza vaccine in this group. Safety monitoring for all three groups is conducted for one month post-vaccination, assessing local symptoms such as redness at the injection site, pain, and systemic symptoms like fever, diarrhoea, weakness, or fatigue. Information related to influenza vaccine effectiveness is obtained by monitoring flu-like syndrome symptoms at months 1, 3, and 6. The researchers also examine interleukin levels, specifically IL-2 and IL-6, before and after vaccination for one month. This examination aims to understand the dynamic changes in both interleukins since IL-2 plays a role in protecting DM patients from influenza virus infections, particularly in preventing secondary infections like pneumonia.

The researcher's hypothesis is that T2DM-CKD patients will exhibit lower antibody responses compared to uncomplicated T2DM patients, and antibody titters against the influenza virus will decline after six months. This study will contribute valuable insights into the frequency of influenza vaccine administration in T2DM and T2DM-CKD groups, potentially reducing morbidity and mortality rates.

ELIGIBILITY:
Inclusion Criteria:

Group 1 (T2DM)

* Individuals with Type 2 Diabetes Mellitus (T2DM)
* Age range: 40-59 years

Group 2 (T2DM-CKD):

* Individuals with Type 2 Diabetes Mellitus (T2DM)
* Age range: 40-59 years
* eGFR (ml/min/1.73 m2) >15
* eGFR (ml/min/1.73 m2) <89
* Proteinuria

Group 3 (Healthy Person) :

* Individuals without Type 2 Diabetes Mellitus (T2DM)
* Age range: 40-59 years

Exclusion Criteria:

* Incomplete medical records
* CKD Stage 5
* Currently pregnant
* Currently on long-term steroid use
* Received influenza vaccine in the last year
* Diagnosed with malignancy
* Autoimmune disease
* History of allergy to chicken eggs or vaccine constituents
* High fever, seizures, or acute infection
* History of COVID infection based on PCR testing with the last PCR result negative <14 days
* History of COVID-19 vaccination <14 days from the last vaccine administration

Ages: 40 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
ILI Morbidity | 6 months
  Determined by the time from treatment to 6 months after
Immunogenicity | 6 months
  Determine the changes in titers over time using the hemagglutination (HA) method at the 1st, 3rd, and 6th months after vaccination.

SECONDARY OUTCOMES:
Inflammatory interleukin measurements | 6 months
  Inflammatory analysis will be performed in the 1st, 3rd, and 6th months.

CONTACTS AND LOCATIONS:
Overall Officials: Nur Atik, MD, Study Chair — Universitas Padjadjaran
Locations (1):
- AMC Hospital, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No